CLINICAL TRIAL: NCT07036029
Title: An Open Label, In-Clinic Study to Assess Respiratory Function and Safety of Escalating Doses of Nalbuphine Extended-Release Tablets (NAL ER) in Subjects With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: NAL ER IPF Respiratory Function and Safety Study
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Trevi Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAL03-101
Record Dates: First submitted 2025-05-29; First posted 2025-06-25 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: nalbuphine
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Nalbuphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- NAL ER (Experimental): Participants will receive 2 doses of placebo (placebo matching NAL ER) over 2 days followed by increasing doses of NAL ER tablets twice daily (BID) over 6 days.
  Interventions: Drug: NAL ER; Drug: Placebo

INTERVENTIONS:
Drug: NAL ER — Oral tablets
  Other Names: Nalbuphine
Drug: Placebo — Oral tablets

SUMMARY:
The primary purpose of this study is to assess the safety and tolerability of escalating doses of NAL ER and to evaluate its effect on respiratory function in participants with IPF.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of IPF as determined by a pulmonologist based on American Thoracic Society (ATS)/ European Respiratory Society (ERS) / Japanese Respiratory Society (JRS) / Asociación Latinoamericana de Tórax (ALAT) guidelines.
* SpO2 ≥ 92%, taken after at least 5 minutes in a sitting position, undisturbed and non-stimulated - Saturation of Hemoglobin with Oxygen as measured by pulse oximetry.
* FVC ≥ 40% of Global Lung Function Initiative (GLI) 2012 predicted values- Forced Vital Capacity, as determined by spirometry adhering to ATS/ERS guidelines.

Exclusion criteria:

* Exacerbation of IPF in the last 3 months.
* Positive results for coronavirus infection (COVID-19) at Day -2, prior to Admission to the clinical research unit (CRU).
* Diagnosis of Chronic Obstructive Pulmonary Disease (COPD), or an forced expiratory volume in 1 second (FEV1)/forced vital capacity (FVC) <0.8.
* Currently using any overnight oxygen therapy at any level or delivered by any modality. Intermittent daytime oxygen use of any duration is allowed.
* Diagnosis of sleep disordered breathing (e.g., sleep apnea).
* Upper or lower respiratory tract infection within the 8 weeks prior to admission to the CRU.
* Clinical history of aspiration pneumonitis.

Note: Other inclusion/exclusion criteria mentioned in the protocol may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Respiratory Function and Safety Assessed by Number of Participants With Increase in End Tidal Partial Pressure of Carbon Dioxide by Capnography (PetCO2) of at Least 10 Millimetres of Mercury (mmHg) From Baseline, or PetCO2>55 mmHg, for at Least 1 Minute | Up to Day 6
Respiratory Function and Safety as Assessed by Number of Participants With a Decrease in Blood Oxygen Saturation (SpO2) to <88% for at Least 1 Minute | Up to Day 6
Respiratory Function and Safety as Assessed by Number of Participants With a Decrease in Respiratory Rate (RR) to <6 Breaths per Minute | Up to Day 6
Safety and Tolerability as Assessed by Number of Participants With Treatment Emergent Adverse Events (TEAEs) | Up to Day 51

CONTACTS AND LOCATIONS:
Overall Officials: Chief Development Officer, Study Director — Trevi Therapeutics
Locations (2):
- Mayo Clinic, Rochester, Minnesota, United States
- Medicines Evaluation Unit Ltd., Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No